CLINICAL TRIAL: NCT01106495
Title: Study of the Effect of EECP on Subclinical Atherosclerosis
Brief Title: Effect of Enhanced External Counterpulsation (EECP) on Subclinical Atherosclerosis
Acronym: SESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yan Zhang, Associate professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EECP-1
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Vascular Endothelium; Counterpulsation, External
MeSH Terms: conditions — Atherosclerosis | interventions — Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External Counterpulsation (Experimental): Enhanced external counterpulsation (EECP) is a noninvasive therapy for the treatment of patients with coronary artery disease.The systolic deflation/diastolic inflation sequence of EECP leads to systolic unloading and diastolic augmentation, resulting in increased blood flow in a pulsatile manner. Patients with subclinical atherosclerosis whose serum LDL high than 160mg/ml receive EECP 1- hour session every working day over a 7 week period. Simvastatin is used to decrease cholesterol level for 7 weeks.
  Interventions: Device: Enhanced External Counterpulsation (EECP); Drug: Simvastatin
- Control (Active Comparator): Subjects whose LDL higher than 160 mg/dl with subclinical atherosclerosis. Simvastatin is used to decrease cholesterol level for 7 weeks.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Device: Enhanced External Counterpulsation (EECP) — EECP one hour per day, 5 hours a week for a total of 35- 36 hours over a 7 week period
  Other Names: EECP
  Arms: Enhanced External Counterpulsation
Drug: Simvastatin — Simvastatin 40 mg/d for 7 weeks as the guideline- driven standard medical treatment
  Other Names: Statin

SUMMARY:
Shear stress maybe the most crucial local factor affecting atherogenesis. The present study investigated the effect of exposure to increased shear stress promoted by Enhanced External Counterpulsation (EECP) on the progression of subclinical atherosclerosis and the underlying inflammation- related molecular mechanisms

DETAILED DESCRIPTION:
Hypercholesterolemic subjects with subclinical atherosclerosis will be randomized into two groups: standard treatment group and standard treatment plus EECP intervention group. The results of ultrasound examination and markers of inflammations will be compared.

ELIGIBILITY:
Inclusion Criteria:

* 20- 70 years old subjects whose LDL higher than 160mg/dl and carotid intima-media thickness higher than 75 percent of his age.

Exclusion Criteria:

* Presence of history of coronary heart disease, stroke or atherosclerotic peripheral disease. Presence of impaired renal function, connective disease, or infectious disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in Intima-media thickness of the carotid artery | 7 weeks
  Change from baseline in Intima-media thickness of the carotid artery measured by Doppler ultrasound equipment at 7 weeks

SECONDARY OUTCOMES:
Change in vascular endothelial function | 7 weeks
  Change from baseline in vascular endothelial function evaluated by flow mediated dilation of the brachial artery
Change in serum markers of inflammation | 7 weeks
  Change from baseline in serum markers of inflammation and laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, MD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat- sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No